CLINICAL TRIAL: NCT00190645
Title: Long-Term Monitoring of Safety in Subjects Treated With Duloxetine for Stress Urinary Incontinence
Brief Title: To Evaluate the Safety of Duloxetine in Patients With Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2688; F1J-MC-SBAW
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
The patients are being followed in this study to determine the safety of taking the medication Duloxetine for a long period of time. The patients participating in this study suffer from Stress Urinary Incontinence.

ELIGIBILITY:
Inclusion Criteria:

Successfully completed the protocol for Study F1J-MC-SBAV.

-

Exclusion Criteria:

Treatment with a drug, not including study medication, that has not received regulatory approval at the time of study entry.

Use of excluded medications within 14 days prior to study entry or at any time during the study.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2001-02; Study Completion 2006-05

PRIMARY OUTCOMES:
To generate long-term safety data for duloxetine in the treatment of women with stress urinary incontinence(SUI).

SECONDARY OUTCOMES:
To collect data to demonstrate the maintenance of effect of duloxetine as measured by Patient Global Impression of Improvement (PGI-I) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Denver, Colorado, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559,1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Oakville, Ontario, Canada